CLINICAL TRIAL: NCT04861974
Title: Estudio Coste-Efectividad "Snapshot" Nacional de Costes robótica vs laparoscópica
Brief Title: Robotic vs Laparoscopic Study. Spanish Cost Effective Snapshot Study
Acronym: ROBOCOSTES
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Benedetto Ielpo, MD, PhD, Hospital del Mar
Other Study IDs: Robocostes
Record Dates: First submitted 2021-04-21; First posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Laparoscopy; Robotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Robotic Distal Pancreatectomy
- Laparoscopic Distal Pancreatectomy
- Robotic Gastrectomy
- Laparoscopic Gastrectomy
- Robotic Funduplication
- Laparoscopic Funduplication
- Robotic Hernioplasty
- Laparoscopic Hernioplasty
- Robotic Rectal Resection
- Laparoscopic Rectal Resection

SUMMARY:
this is a prospective no randomized study of cost effectiveness of laparoscopic vs robotic study of Distal pancreatectomy, Hernioplasty for inguinal hernia and Rectal resection

DETAILED DESCRIPTION:
Robotic is having increased interest in the last decade and on of its limits is the cost.

From previous report Robotic surgery entails higher costs. However, cost solely is not enough to validate a new procedure. Whenever a new technology is introduced it is important to evaluate cost and improved quality of life as well, which is the Cost Effectiveness (CE) study.

The aim of our study is to evaluate in Spain the CE of laparoscopic and robotic procedure of Distal Pancreatectomy, Gastrectomy, Nissen procedure, Rectal resection and Inguinal hernia repair.

This is a prospective snapshot study during 6 months in which patients are included from several Spanish centers. Cost are defined according to the spain official cost data recorded from the RECH (https://www.rechosp.org).

Main clinical outcomes are gathered divided in intra operative and post operative data.

Quality of life (EQ 5D-5L) is recorded as well pre operatively and post operatively at 30 days and 9 days from the surgery, time in which the follow up is ended.

A cost effectiveness analysis is finally performed:

A model-based cost-utility analysis estimating mean costs and QALYs per patient was performed.

The Institute for Validation of Clinical Efficacy (IVEC) of the HM Hospitals group was responsible for capturing costs ascribed to each patient's treatment. The total direct hospital costs of care, with the exception of the acquisition or maintenance of the robotic device.

Materials and medicines used during surgery were standardized so that the same materials were used in all patients undergoing surgery regardless of the technique employed (Robotic or Laparoscopic). Operative costs included the cost of the operating room in relation to the operative time, and all required supplies (including all laparoscopic devices, sutures, and instruments), anaesthesia, laboratory and related blood transfusion costs when required. Hospitalization costs included costs associated with room and board, the length of hospital stay (including intensive care, medications, blood transfusion, parenteral nutrition and radiology charge) and costs for surgical visits (programmed and emergency) as well as readmission costs up to 90 days from surgery. The direct costs of the professionals involved have not been calculated as they did not vary between the two types of operation. A discount rate of 3% per year is used in the estimation of the costs and QALYs, as recommended by health economic guidelines (9) All costs are presented in Euros (exchange rate 2021).

Stochastic cost-utility analysis was undertaken, whereby the incremental cost-effectiveness ratio (ICER) was estimated using overall costs of the RRR and LRR procedures and QALYs derived from patient interviews, in order to find the incremental cost per QALYs gained.

Net monetary benefits (NMBs) were calculated in order to estimate the maximum willingness to pay (WTP) of decision makers for a QALY gained. The NMB was calculated as the mean QALYs per patient multiplied by WTP threshold minus the mean cost per patient for the treatment. The decision rule is to adopt the treatment if the NMB > 0, and the alternative with the highest NMB represents best value for money.

Sensitivity analysis A sensitivity analysis was carried out in order to propagate the uncertainty of the estimations to the results of the model. We used a multivariate and stochastic sensitivity analysis performed by 5,000 Monte Carlo simulations. The cost-effectiveness plane was used to represent all pairs of solutions of the model.

The results of the one-way sensitivity analysis are shown in the tornado diagram which depicts graphically how variations in each input affect the outcome. The 95% confidence intervals around the base case values were derived using the 2.5 and 97.5 percentiles calculated from the sensitivity analysis.

The tornado diagram is stacked in order of decreasing width, indicating that variations in inputs near the top (Total Costs Robotic) have the greatest effect on the outcome, while variations in inputs near the bottom (QALYs discount rate) have relatively small effects on the outcome.

Acceptability curve The investigators also computed a cost-effectiveness acceptability curve which plots the probability that the Robotic was cost-effective relative to Laparoscopy over a reasonable range of levels of willingness-to-pay.

Although in Spain there is no specific willing to pay threshold in healthcare, according to the National Institute for Health Care Excellence (NICE), the investigators used a willingness-to-pay of 20,000 € and 30,000 € per QALY as a threshold to recognize which treatment was most cost-effective

Statistics Data have been recorded in a SPSS Statistics Version 20.0 database and are expressed as median values (interquartile range-IQR 25-75). Categorical data are presented as numbers (%). To compare the means of the quantitative variables when the variables followed a normal distribution, a variance analysis and a Student's t-test were used. For the rest of the variables, both Mann-Whitney and Kruskal-Wallis tests were performed. Cost, QALYs and incremental results are presented in a 95% Confidence Interval. A p value < .05 was considered significant. Data herein reported are for patients who reached a minimum of one year of follow up.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery with indication of distal Pancreatectomy , Gastrectomy, Hernioplasty, Rectal resection and Nissen performed by laparoscopy or robotic
* >18 years old

Exclusion Criteria:

* Patients who do not want to participate
* Previous abdominal surgeries

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Elective surgery with indication of distal Pancreatectomy , Gastrectomy, Hernioplasty, Rectal resection and Nissen
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-06-15 (Estimated); Primary Completion 2022-04-15 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
Cost Effectiveness | 90 days
  This is the increased cost differences of the new technology to improve the quality of life after the intervention